CLINICAL TRIAL: NCT05317312
Title: A Randomized, Double Blind, Placebo Controlled, Parallel Group, Dose Response Study of MR-107A-02 in the Treatment of Post Surgical Dental Pain.
Brief Title: Study of MR-107A-02 in the Treatment of Post Surgical Dental Pain.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mylan Specialty, LP (Industry)
Responsible Party: Sponsor
Organization: Viatris Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MELO-TFZ-2001
Record Dates: First submitted 2022-03-16; First posted 2022-04-07 (Actual); Results first posted 2023-08-07 (Actual); Last update posted 2023-08-07 (Actual); Status verified 2023-08

CONDITIONS: Acute Pain; Post Operative Pain; Pain
MeSH Terms: conditions — Acute Pain; Pain, Postoperative; Pain

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: double blind, placebo controlled
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- MR-107A-02 1.25 mg twice in a 24 hour period (Experimental): Oral tablet, one day of dosing
  Interventions: Drug: MR-107A-02
- MR-107A-02 5 mg twice in a 24 hour period (Experimental): Oral tablet, one day of dosing
  Interventions: Drug: MR-107A-02
- MR-107A-02 15 mg twice in a 24 hour period (Experimental): Oral tablet, one day of dosing
  Interventions: Drug: MR-107A-02
- Placebo twice in a 24 hour period (Placebo Comparator): Oral tablet, one day of dosing
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MR-107A-02 — MR-107A-02 oral tablet
  Arms: MR-107A-02 1.25 mg twice in a 24 hour period; MR-107A-02 15 mg twice in a 24 hour period; MR-107A-02 5 mg twice in a 24 hour period
Drug: Placebo — Placebo oral tablet
  Arms: Placebo twice in a 24 hour period

SUMMARY:
MR-107A-02 is being studied to investigate its efficacy, safety and dose-response after dental surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females ≥18 years of age.
2. Requirement for dental surgery for extraction of ≥2 third molars, at least 1 of which involves partial or complete mandibular bony impaction.
3. Pain Intensity (PI) using a Numeric Pain Rating Scale (NPRS) ≥5 during the 5 hours following the end of surgery in the eligibility assessment as well as in the baseline assessment immediately pre-dosing.
4. Rating of moderate or severe pain on a 4-point categorical pain rating scale (i.e., none, mild, moderate, severe) during the 5 hours following the end of surgery.

Exclusion Criteria:

1. Previously dosed with MR-107A-02.
2. Subject with known hypersensitivity to nonsteroidal anti-inflammatory drugs (NSAIDs).
3. Active GI bleeding or a history of peptic ulcer disease, active inflammatory bowel disease, e.g., Crohn's Disease or ulcerative colitis,or bleeding disorders that may affect coagulation.
4. Moderate or severe hypertension, prior stroke or transient ischemic attack.
5. Use of any investigational drug within 28 days, or 5 half-lives, prior to consent whichever is longer.
6. Use of medications with the potential to interact with MR-107A-02.
7. Other acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2022-03-31 (Actual); Primary Completion 2022-06-15 (Actual); Study Completion 2022-06-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Research Facility 201, Salt Lake City, Utah, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 111 subjects were enrolled / randomized but only 110 subjects were treated.
Period: Overall Study
Arm/Group | MR-107A-02 1.25 mg Twice in a 24 Hour Period | MR-107A-02 5 mg Twice in a 24 Hour Period | MR-107A-02 15 mg Twice in a 24 Hour Period | Placebo Twice in a 24 Hour Period
Started | 28 | 28 | 27 | 27
Completed | 28 | 27 | 26 | 26
Not Completed | 0 | 1 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1
Not completed — Excluded as exclusion criteria was met. | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MR-107A-02 1.25 mg Twice in a 24 Hour Period | MR-107A-02 5 mg Twice in a 24 Hour Period | MR-107A-02 15 mg Twice in a 24 Hour Period | Placebo Twice in a 24 Hour Period | Total
Number analyzed (Participants) | 28 | 28 | 27 | 27 | 110
Age, Continuous [Mean (Standard Deviation); unit: years] | 18.9 (1.45) | 19 (1.52) | 19.3 (1.94) | 18.7 (1.13) | 19 (1.53)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 16 | 16 | 14 | 63
  Male | 11 | 12 | 11 | 13 | 47
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 4 | 2 | 4 | 12
  Not Hispanic or Latino | 26 | 24 | 25 | 23 | 98
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 28 | 28 | 27 | 27 | 110

OUTCOME MEASURES:

1. Primary Outcome: Overall Summed Pain Intensity Difference (SPID)
Description: Participants assessed Pain Intensity (PI) using a 0-10 numeric pain rating scale (NPRS) where 0 is no pain and 10 is worst pain imaginable. PI was assessed 18 times within 24 hours after the first study dose, and immediately before any rescue medication and/or at early termination. The participant's baseline PI was subtracted from the timepoint PI, to derive a Pain Intensity Difference (PID) for each timepoint. Overall Summed Pain Intensity Difference (SPID) measures pain intensity change relative to baseline over the 24 hour period after dosing, and corresponds to the Area Under the Curve (AUC) of the PID. In this study, higher positive Overall SPID indicates better pain improvement. Overall SPID could range from -120 to 240. Two hour windowed last observation carried forward was used as applicable where PI score obtained before a rescue medication replaced PI score for each timepoint within 2 hours following rescue dose.
Time Frame: 24 hours after the first dose
Population: Modified Intent-to-treat Analysis Set
Measure: Mean (Standard Deviation); unit: score on a scale x hours
Arm/Group | MR-107A-02 1.25 mg Twice in a 24 Hour Period | MR-107A-02 5 mg Twice in a 24 Hour Period | MR-107A-02 15 mg Twice in a 24 Hour Period | Placebo Twice in a 24 Hour Period
Number analyzed (Participants) | 28 | 28 | 27 | 27
score on a scale x hours | 74.5 (46.49) | 82.4 (37.78) | 96.8 (35.31) | 50.5 (37.26)
Statistical Analysis 1: Comparison: MR-107A-02 1.25 mg Twice in a 24 Hour Period vs Placebo Twice in a 24 Hour Period; Test type: Superiority; p = 0.123, Emax; Mean Difference (Final Values) = 18.7, 95% CI 2-sided [-5.2 to 42.7], Standard Error of Mean 12.08 — The estimated difference between 1.25mg bid and placebo is based on the Emax model. The values that appear in the Outcome Measure Data Table are observed values
Statistical Analysis 2: Comparison: MR-107A-02 5 mg Twice in a 24 Hour Period vs Placebo Twice in a 24 Hour Period; Test type: Superiority; p < 0.001, Emax; Mean Difference (Final Values) = 34.7, 95% CI 2-sided [14.4 to 55.0], Standard Error of Mean 10.25; The estimated difference between 5mg bid and placebo is based on the Emax model. The values that appear in the Outcome Measure Data Table are observed values
Statistical Analysis 3: Comparison: MR-107A-02 15 mg Twice in a 24 Hour Period vs Placebo Twice in a 24 Hour Period; Test type: Superiority; p < 0.001, Emax; Mean Difference (Final Values) = 42.8, 95% CI 2-sided [23.9 to 61.7], Standard Error of Mean 9.53 — The estimated difference between 15mg bid and placebo is based on the Emax model. The values that appear in the Outcome Measure Data Table are observed values

2. Secondary Outcome: Pain Intensity Using a Number Pain Rating Scale Utilizing 6-hour Windowed Last Observation Carried Forward (W6LOCF)
Description: 10 point scale, where 0 is no pain and 10 is the worst pain imaginable; 6-hour windowed last observation carried forward (W6LOCF) utilizes "pain right now" just prior to rescue medication use and censors subsequent pain intensity values for 6 hours when calculating SPIDs
Time Frame: 24 hours after first dose
Population: Modified Intent-to-treat Analysis Set
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MR-107A-02 1.25 mg Twice in a 24 Hour Period | MR-107A-02 5 mg Twice in a 24 Hour Period | MR-107A-02 15 mg Twice in a 24 Hour Period | Placebo Twice in a 24 Hour Period
Number analyzed (Participants) | 28 | 27 | 27 | 27
score on a scale | 2.5 (1.88) | 3.1 (2.32) | 2.4 (1.72) | 3.5 (2.29)
Statistical Analysis 1: Comparison: MR-107A-02 1.25 mg Twice in a 24 Hour Period vs Placebo Twice in a 24 Hour Period; Test type: Superiority; Mean Difference (Final Values) = -0.9, 95% CI 2-sided [-2.0 to 0.2], Standard Error of Mean 0.56 — The estimated difference between 1.5mg bid and placebo is based on Mixed Model Repeated Measures.The values in the Outcome Measure Data are observed mean values
Statistical Analysis 2: Comparison: MR-107A-02 5 mg Twice in a 24 Hour Period vs Placebo Twice in a 24 Hour Period; Test type: Superiority; Mean Difference (Final Values) = -0.7, 95% CI 2-sided [-1.8 to 0.4], Standard Error of Mean 0.56 — The estimated difference between 5mg bid and placebo is based on Mixed Model Repeated Measures. The values in the Outcome Measure Data are observed mean values
Statistical Analysis 3: Comparison: MR-107A-02 15 mg Twice in a 24 Hour Period vs Placebo Twice in a 24 Hour Period; Test type: Superiority; Mean Difference (Final Values) = -0.8, 95% CI 2-sided [-1.9 to 0.3], Standard Error of Mean 0.56 — The estimated difference between 15mg bid and placebo is based on Mixed Model Repeated Measures.. The values in the Outcome Measure Data are observed mean values

3. Secondary Outcome: Time to Perceptible Pain Relief.
Description: Measured by double stopwatch technique. The time to onset of first perceptible relief (time that the first watch is stopped) is defined as the postdose time at which the subject first begins to feel pain relief at their estimation.
Time Frame: 24 hours after first dose
Population: Modified Intent-to-treat Analysis Set
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | MR-107A-02 1.25 mg Twice in a 24 Hour Period | MR-107A-02 5 mg Twice in a 24 Hour Period | MR-107A-02 15 mg Twice in a 24 Hour Period | Placebo Twice in a 24 Hour Period
Number analyzed (Participants) | 21 | 21 | 26 | 10
hours | 0.9 [0.6 to 3.4] | 0.7 [0.5 to 0.9] | 0.6 [0.4 to 0.7] | NA [0.8 to NA] — Values marked NA (not applicable) have insufficient counts of events to be estimable from the K-M methodology.
Statistical Analysis 1: Comparison: MR-107A-02 1.25 mg Twice in a 24 Hour Period vs Placebo Twice in a 24 Hour Period; Test type: Superiority; p = 0.036, Log Rank
Statistical Analysis 2: Comparison: MR-107A-02 5 mg Twice in a 24 Hour Period vs Placebo Twice in a 24 Hour Period; Test type: Superiority; p = 0.006, Log Rank
Statistical Analysis 3: Comparison: MR-107A-02 15 mg Twice in a 24 Hour Period vs Placebo Twice in a 24 Hour Period; Test type: Superiority; p < 0.001, Log Rank

4. Secondary Outcome: Time to Meaningful Pain Relief
Description: Measured by double stopwatch technique The time to meaningful pain relief (time that the second watch is stopped) is defined as the postdose time at which the subject begins to feel meaningful pain relief at their estimation
Time Frame: 24 hours after first dose
Population: Modified Intent-to-treat Analysis Set
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | MR-107A-02 1.25 mg Twice in a 24 Hour Period | MR-107A-02 5 mg Twice in a 24 Hour Period | MR-107A-02 15 mg Twice in a 24 Hour Period | Placebo Twice in a 24 Hour Period
Number analyzed (Participants) | 14 | 13 | 21 | 6
hours | 4.5 [3.0 to 6.8] | 5.0 [1.5 to NA] — Values marked NA (not applicable) have insufficient counts of events to be estimable from the K-M methodology. | 1.5 [1.0 to 2.3] | 3.9 [2.9 to NA] — Values marked NA (not applicable) have insufficient counts of events to be estimable from the K-M methodology.
Statistical Analysis 1: Comparison: MR-107A-02 1.25 mg Twice in a 24 Hour Period vs Placebo Twice in a 24 Hour Period; Test type: Superiority; p = 0.411, Log Rank
Statistical Analysis 2: Comparison: MR-107A-02 5 mg Twice in a 24 Hour Period vs Placebo Twice in a 24 Hour Period; Test type: Superiority; p = 0.383, Log Rank
Statistical Analysis 3: Comparison: MR-107A-02 15 mg Twice in a 24 Hour Period vs Placebo Twice in a 24 Hour Period; Test type: Superiority; p < 0.001, Log Rank

5. Secondary Outcome: Patient's Global Assessment of Pain Control
Description: 5 point PGA (Patient's Global Assessment) of pain control scale, where 0 is poor, 1 is fair, 2 is good, 3 is very good, and 4 is excellent
  Responder = 2 is good, 3 is very good, and 4 is excellent Non-responder = 1 is fair, 0 is poor, and missing values.
Time Frame: 24 hours
Population: Subjects reporting a PGA score of 2 (good) or better defined as a responder
Measure: Number; unit: percentage of PGA responders
Arm/Group | MR-107A-02 1.25 mg Twice in a 24 Hour Period | MR-107A-02 5 mg Twice in a 24 Hour Period | MR-107A-02 15 mg Twice in a 24 Hour Period | Placebo Twice in a 24 Hour Period
Number analyzed (Participants) | 28 | 28 | 27 | 27
percentage of PGA responders | 60.7 | 67.9 | 85.2 | 33.3
Statistical Analysis 1: Comparison: MR-107A-02 1.25 mg Twice in a 24 Hour Period vs Placebo Twice in a 24 Hour Period; Test type: Superiority; p = 0.042, Chi-squared; Risk Difference (RD) = 27.4, 95% CI 2-sided [2.0 to 52.7]
Statistical Analysis 2: Comparison: MR-107A-02 5 mg Twice in a 24 Hour Period vs Placebo Twice in a 24 Hour Period; Test type: Superiority; p = 0.01, Chi-squared; Risk Difference (RD) = 34.5, 95% CI 2-sided [9.7 to 59.3]
Statistical Analysis 3: Comparison: MR-107A-02 15 mg Twice in a 24 Hour Period vs Placebo Twice in a 24 Hour Period; Test type: Superiority; p < 0.001, Chi-squared; Risk Difference (RD) = 51.9, 95% CI 2-sided [29.6 to 74.1]

6. Secondary Outcome: Rescue Medication Use
Description: Percentage of subjects using rescue medication from 0-24 hours
Time Frame: 24 hours after first dose
Population: Rescue Medication Used within 24h
Measure: Number; unit: percentage of participants
Arm/Group | MR-107A-02 1.25 mg Twice in a 24 Hour Period | MR-107A-02 5 mg Twice in a 24 Hour Period | MR-107A-02 15 mg Twice in a 24 Hour Period | Placebo Twice in a 24 Hour Period
Number analyzed (Participants) | 28 | 28 | 27 | 27
percentage of participants | 42.9 | 57.1 | 29.6 | 74.1
Statistical Analysis 1: Comparison: MR-107A-02 1.25 mg Twice in a 24 Hour Period vs Placebo Twice in a 24 Hour Period; Test type: Superiority; p = 0.019, Chi-squared; Risk Difference (RD) = -31.2, 95% CI 2-sided [-55.9 to -6.5]
Statistical Analysis 2: Comparison: MR-107A-02 5 mg Twice in a 24 Hour Period vs Placebo Twice in a 24 Hour Period; Test type: Superiority; p = 0.187, Chi-squared; Risk Difference (RD) = -16.9, 95% CI 2-sided [-41.6 to 7.8]
Statistical Analysis 3: Comparison: MR-107A-02 15 mg Twice in a 24 Hour Period vs Placebo Twice in a 24 Hour Period; Test type: Superiority; p = 0.001, Chi-squared; Risk Difference (RD) = -44.4, 95% CI 2-sided [-68.3 to 20.6]

ADVERSE EVENTS:
Time Frame: Study period reporting of Adverse Events was up to 7 days post first dose. Subjects were reminded that AEs should be reported to the study staff up to 30 days after the last dose of study medication.
Description: An adverse event is any untoward medical occurrence in a patient/ clinical investigation subject administered a pharmaceutical product and which does not necessarily have to have a causal relationship with treatment.
  An adverse event can therefore be any unfavorable and unintended sign (including an abnormal laboratory/ physical findings, symptom, or disease (new/ exacerbated) temporally associated with the use of a medicinal product whether or not considered related to the medicinal product.
Arm/Group | MR-107A-02 1.25 mg Twice in a 24 Hour Period | MR-107A-02 5 mg Twice in a 24 Hour Period | MR-107A-02 15 mg Twice in a 24 Hour Period | Placebo Twice in a 24 Hour Period
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/28 | 0/27 | 0/27
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/28 | 0/27 | 0/27
Other Adverse Events (participants affected / at risk) | 3/28 | 7/28 | 8/27 | 8/27
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | MR-107A-02 1.25 mg Twice in a 24 Hour Period (N=28) | MR-107A-02 5 mg Twice in a 24 Hour Period (N=28) | MR-107A-02 15 mg Twice in a 24 Hour Period (N=27) | Placebo Twice in a 24 Hour Period (N=27)
Nausea (Gastrointestinal disorders) | 1 | 5 | 2 | 2
Vomitting (Gastrointestinal disorders) | 0 | 0 | 2 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Blood bilirubin increased (Investigations) | 2 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 2 | 3
Dizziness (Nervous system disorders) | 0 | 1 | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Subject to a multi-site coordination for publication, Institution and Investigator may publish its results by providing a copy of any presentation/publication derived from the Study for review and comment at least 30 days in advance of any disclosure, presentation, or submission for publication in order for the removal of anything that Sponsor identifies as trade secrets, proprietary information or Confidential Information.

DOCUMENTS (2):
  • Study Protocol (2022-02-15): https://cdn.clinicaltrials.gov/large-docs/12/NCT05317312/Prot_000.pdf
  • Statistical Analysis Plan (2022-07-23): https://cdn.clinicaltrials.gov/large-docs/12/NCT05317312/SAP_001.pdf